CLINICAL TRIAL: NCT07250646
Title: A Phase 1 Study of Rebecsinib, a Spliceosome Modulator That Inhibits ADAR1, in Patients With Relapsed or Refractory Secondary Acute Myeloid Leukemia or Higher-Risk Myelofibrosis
Brief Title: A Study of Rebecsinib for Patients With Relapsed/Refractory Secondary Acute Myeloid Leukemia or High Risk Myelofibrosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspera Biomedicines, Inc. (Industry)
Collaborators: Tempus AI (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASPE-01-01
Record Dates: First submitted 2025-08-01; First posted 2025-11-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Secondary AML; Myelofibrosis
Keywords: sAML; MF
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Intervention Model Description: This study includes a Modified Fibonacci design of up to 11- dose cohorts until an MTD or biologically active dose is reached or any participant experiences a ≥Grade 2 AE. An accelerated dose escalation with 1 patient per dose will be performed at doses of 0.2, 0.4, 0.6, and 0.8 mg/kg.
  At a dose level of 1.0 mg/kg or at a dose where a grade 2 or greater adverse event occurs, a 3+3 design escalation will be performed with doses of 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 mg/kg with an expansion cohort of 3 patients at the MTD, so that a total of 6 patients will be evaluable at the MTD with an extra 3 patients added if RP2D is lower than MTD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: rebecsinib — Rebecsinib is administered by intravenous infusion on Days 1, 4, 8, and 11 of the 28 day cycle. Doses to be tested are 0.2, 0.4, 0.6, 0.8, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, and 8.0 mg/kg based in ideal body weight (IBW).
  Other Names: 17S-FD-895

SUMMARY:
The purpose of this study is to test the safest and most effective dose of a new investigational drug, rebecsinib. Participants in this study will have either Secondary Acute Myeloid Leukemia (sAML) that has either returned (relapsed) or not responded to treatment (refractory) or have higher risk Myelofibrosis (MF). Participants will receive a study drug infusion on Day 1, Day 4, Day 8 and Day 11 of each 28-day cycle for a total of 6 cycles.

DETAILED DESCRIPTION:
The primary objective is to determine the maximum tolerated dose or biologically active dose of rebecsinib when given on days 1, 4, 8, and 11 of each 28 days cycle to patients with relapsed or refractory secondary acute myeloid leukemia (sAML), who have evolved from Myelodysplastic Syndrome (MDS) or myeloproliferative neoplasms (MPNs), or patients with higher-risk myelofibrosis. The other primary objective is to determine the safety and tolerability of rebecsinib by ongoing evaluation of adverse events (AEs), as assessed according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0).

Study outcomes will be measured by adverse event data, response rates, progression free survival and overall survival. Pharmacodynamics and plasma pharmacokinetics of rebecsinib will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent.
2. Must have a refractory myeloid neoplasm (5th Edition WHO Classification of Tumors) consisting of secondary AML (sAML), which has evolved from antecedent MDS, MPN, MDS/MPN, or have higher-risk MF defined by DIPSS Plus or MIPSS70+ version 2.0, and excess bone marrow blasts (> 5%). Patients with sAML, defined as AML with an antecedent history of MDS or MPN or WHO AML with myelodysplasia related genetic changes or WHO AML with myelodysplasia related cytogenetic abnormalities. Must be ineligible for bone marrow transplantation at the time of enrollment and have relapsed or be refractory or intolerant to available therapies, such as anthracycline chemotherapy, epigenetic modifier therapy (azacytidine or decitabine) or venetoclax including any treatment that is active in specific mutations if relevant (e.g., FLT3 inhibitors for patients with FLT3 mutations). If the patient has not received intensive induction chemotherapy in the past as a result of being unfit for chemotherapy, then the patient must have undergone at least one line of epigenetic modifier or other available therapy. If the patient has received intensive induction therapy, then the patient must have undergone at least two lines of therapy. If a patient has a FLT3 or IDH mutation, prior therapy must include a FLT3 or an IDH inhibitor. Relapse is defined as the recurrence of excess leukemic blasts in the marrow after previously achieving a complete remission, or complete remission with incomplete count recovery. Refractory refers to persistent excess leukemic blasts after two cycles of standard anthracycline containing induction, or one cycle of a high dose cytarabine containing regimen, or one cycle of a non-intensive regimen.
3. Calculated Creatinine clearance (CrCl) > 60 mL/min (based upon the Cockcroft- Gault Equation [CrCl = (140-age) * ideal body wt (in kg) * (0.85 if female) / (72 * Cr)]. Estimate Ideal body weight in (kg) Males: IBW = 50 kg + 2.3 kg for each inch over 5 feet. Females: IBW = 45.5 kg + 2.3 kg for each inch over 5 feet.
4. Has recovered from the toxic effects of prior therapy to their clinical baseline.
5. Subjects must be aged 18 years or older.
6. Both men and women of all races and ethnic groups are eligible for this trial.
7. Women of childbearing potential (not postmenopausal for at least one year or not surgically incapable of bearing children) must agree not to become pregnant for the duration of the study. Both men and women must agree to use a barrier method of contraception for the duration of the study and until 10 weeks after the final dose of rebecsinib.
8. Women of child-bearing potentialmust have a negative serum or urine pregnancy test.
9. For sAML and high risk MF, at relapse must have ≥5% leukemic bone marrow blasts.
10. Subjects must have an ECOG performance status of 0-2.
11. Hemoglobin ≥ 8.0 g/dL. This is to alleviate immediate concomitant need for transfusion via institutional guidelines for transfusion for symptomatic anemia.
12. Total bilirubin ≤ 1.5 times upper limit of normal.
13. ALT and AST ≤ 1.5 times upper limit of normal
14. Prothrombin time international normalized ratio (INR) ≤ 2; AND Partial thromboplastin time ≤ 1.66 times upper limit of normal.

Exclusion Criteria:

1. Pregnant or breast feeding females are excluded.
2. Previous hematopoietic cell transplant.
3. Patients who are currently receiving another investigational agent are excluded.
4. Patients who have had chemotherapy (e.g., HMA therapy, chemotherapy, immunotherapy) or participation in any investigational drug treatment within 2 weeks or 5-half lives, whichever is more, of initiation of rebecsinib or at any time during the study.
5. Current infection requiring systemic antibiotics.
6. Active infection with HIV, HBV, or HCV.
7. Concurrent malignancy or prior malignancy within the previous 3 years (other than completely resected carcinoma in situ or localized non-melanoma skin cancer).
8. Known central nervous system (CNS) involvement by malignancy.
9. Untreated autoimmunity such as autoimmune hemolytic anemia or immune thrombocytopenia.
10. Known uncompensated hypothyroidism (defined as TSH greater than 2x upper limit of normal not treated with replacement hormone).
11. Insufficient recovery from surgery-related wound healing.
12. Impaired cardiac function including any of the following:

    1. Myocardial infarction within 6 months of starting study drug;
    2. A past medical history of clinically significant ECG abnormalities, including QTc 470 msec or greater.
    3. Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
13. A QT ->470 msec on ECG.
14. On medication that is an inducer or inhibitor of CYP3A4, CYP2C9, CYP2C19, CYP2B6 and hepatic uptake transporters (e.g. OATP1B1/3, OAT1/2 OCT 1/2), or is metabolized by CYP2C9, 2C19, and 2B6. If they are an inducer or inhibitor or a known substrate of CYP2B6, CYP2C9, and CYP2C19 where minimal changes in drug concentration may lead to serious adverse reactions, the drug should be withdrawn for a minimum of 5 half lives or particular attention should be paid to toxicities or appropriate dose modifications to these drugs made.
15. Patients who in the opinion of the investigator may be unable to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose | From first dose through 28 days after initial dose for dose all finding cohorts, approximately 2 years.
  Find the rate of dose limiting toxicities (DLTs) to establish the maximum tolerated dose (MTD) or biologically active dose of rebecsinib when given on days 1, 4, 8, and 11 of each 28 days cycle.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From enrollment to initiation of new therapy for each subject, approximately 4 months.
  To determine the safety and tolerability of rebecsinib by ongoing evaluation of treatment-emergent adverse events (AEs) by collecting description, timing, grade [CTCAE v5.0], severity, seriousness, and relatedness of all events.

SECONDARY OUTCOMES:
Assess Clinical Activity through Overall Response Rate using 2017 ELN Response Criteria | From enrollment through disease assessment that shows progression, approximately 4 months.
  To assess clinical activity by evaluating overall response rate. Overall Response Rate (ORR): Percentage of patients achieving Complete Remission (CR) + Partial Remission (PR) as defined by the revised 2017 ELN response criteria for AML
Assess Clinical Activity through Duration of Response | From enrollment through disease assessment that shows progression, approximately 4 months
  To assess clinical activity by evaluating duration of response. Duration of response is defined as number of days from day of complete or partial remission to day of relapse
Assess Clinical Activity through Progression Free Survival Using 2017 ELN Response Criteria | From enrollment through disease assessment that shows progression, approximately 4 months
  To assess clinical activity by evaluating progression free survival, defined by the revised 2017 ELN response criteria for AML
Assess Clinical Activity through Overall Survival using the revised 2017 ELN response criteria for AML | From enrollment through disease assessment that shows progression, approximately 4 months
  To assess clinical activity by evaluating overall survival, defined by the revised 2017 ELN response criteria for AML

CONTACTS AND LOCATIONS:
Overall Officials: James Mangan, MD, PhD, Principal Investigator — UC San Diego Moores Cancer Center
Locations (1):
- UC San Diego Moores Cancer Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided